CLINICAL TRIAL: NCT04372537
Title: Medical Hypnosis Against Anxiety and Pain in Electro-neuro-myography
Acronym: HYPNOMADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019_42; 2020-A00092-37 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Anxiety
Keywords: hypnosis; electro-neuro-myography; anxiety; pain; analgesia
MeSH Terms: conditions — Anxiety Disorders; Pain; Agnosia | interventions — Hypnosis; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental): Patients will benefit from formal hypnosis (trance induction, hypno analgesia, comfort suggestions) and/or conversational hypnosis (confusion, distraction, use of chosen words, goodwill using verbal and non verbal languages).
  They will also get to be informed of the proceedings of the performed examination as the standard procedure group.
  Interventions: Behavioral: hypnosis
- Standard procedure group. (Active Comparator): Patients will be informed of the proceedings of the performed examination, without using any hypnosis technique.
  This corresponds to the standard clinical procedures used while performing an electroneuromyogram.
  Interventions: Behavioral: standard care

INTERVENTIONS:
Behavioral: hypnosis — use of hypnosis.
  Arms: Hypnosis
Behavioral: standard care — standard clinical procedure
  Arms: Standard procedure group.

SUMMARY:
Electroneuromyography (ENMG) is a regular neurological investigation that might be painful or unpleasant. Medical hypnosis can avoid these sensations, and is more and more performed during other medico-technical procedures (radiology, biopsies for example). This study aims at evaluate the effect of medical hypnosis on pain and anxiety during ENMG, in patients presenting with anxiety. Our hypothesis is that the anxiety and pain during ENMG will be lower in patients with hypnosis compared to patients with standard care. This will allow us to help patients with this tool during most ENMG procedures, and extend it to other electrophysiological procedures in the future.

DETAILED DESCRIPTION:
Medical hypnosis is more and more used during some medico-technical investigational procedures, such as interventional radiology, dental procedures, baby deliveries. Using the modified conscious state induced by trance or by conversational hypnosis (thanks to verbal and nonverbal language) allows a better tolerance of these procedures. Only very few situations recommend against this approach.

ENMG is a frequently performed procedure in neurology to explore neuromuscular functions. It implies electric stimulations, needle insertion and needs the patient cooperation and the patient's well-being. This is all the more necessary that this procedure may be repeated for a patient along his/her life.

Only one study evaluated the effect of hypnosis on pain and anxiety during ENMG (Slack and al., 2009). Despite a low statistical power due to a small sample, it showed a reduction of the maximal pain during the needle electromyography.

More proof is therefore needed to assess the efficacity of hypnosis against pain and anxiety during ENMG.

Several members of our nurse and medical team have an experience in hypnosis practice and this procedure is sometimes used in some patients, when specifically required, alone or with other analgesic procedures (like nitrous oxide), but not in the current standard practice. This is mainly useful in patients with anxiety.

This study's principal objective is then to evaluate the effect of an hypnosis procedure, compared to a standard clinical procedure alone, on pain consecutive to ENMG, in patients presenting with anxiety when attending an ENMG. The secondary objective is to assess the effect of hypnosis on anxiety consecutive to the ENMG.

This is a monocentric, controlled, randomized, open-labeled study, with two balanced arms. The study cannot be blind since the members of the staff will apply at the same time the hypnosis procedures and the ENMG investigations.

Patients who have to undergo an ENMG due to their standard care investigations will be consecutively included as long as they're taken care of by members of the staff with an hypnosis experience and express any anxiety.

48 patients in each group will have to be include to achieve a sufficient power.

Statistical analyses will be blindly performed by our methodology, biostatistics and data management unit. All tests will be bilateral with an alpha risk of 5%, with an intention-to-treat procedure.

Our hypothesis is a reduction of pain and anxiety in the hypnosis group compared to the standard care one.

If this is confirmed, it will be an argument to offer this procedure in a systematic way to any patient with anxiety who has to undergo an ENMG as well as developing its use in other electrophysiological investigations.

ELIGIBILITY:
Inclusion Criteria:

* patient admitted for ENMG manifesting: spontaneous verbal anxiety about taking the test/- a state of anxiety about the examination, as evidenced by a dark colour on a wellness scale used in the unit
* with a good understanding of the French language
* able to complete self-questionnaires
* Patient who has given written consent to participate in the trial
* Socially insured patient

Exclusion Criteria:

* algesic sensitivity disorders
* known history of psychiatric illness or current known psychiatric illness: severe depression, psychosis
* Administrative reasons: inability to receive informed information, inability to participate in the entire study, lack of social security coverage, refusal to sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Pain score evaluated by analogue visual scale | at the end of electro-neuro-myography exam
  EVA measures the intensity of pain on a scale of 0 (no pain) to 10 (maximum pain imaginable)

SECONDARY OUTCOMES:
Anxiety score evaluated by analogue visual scale | at the end of electro-neuro-myography exam
  EVA measures the intensity of anxiety on a scale of 0 (calm) to 10 (maximum anxiety)
anxiety score evolution evaluated by analogue visual scale | between baseline and at the end of electro-neuro-myography exam
  Anxiety evolution pre/post electro-neuro-myography exam (EVA measures the intensity of anxiety on a scale of 0 (calm) to 10 (maximum anxiety imaginable) will be compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Perrine Bocquillon, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France